CLINICAL TRIAL: NCT01672424
Title: Ultrasound Assessment of Gastric Emptying Following the Addition of a High Protein Drink vs Ice Chips During Labor
Brief Title: Ultrasound Assessment of Gastric Emptying
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO11090441
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Pregnancy
Keywords: NPO; Gastric Emptying; Ice Chips; Protein Drink; Ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group P: High Protein Drink: Patients receiving the high protein drink with 30 grams of protein in 11 fluid ounces.
  Interventions: Other: Protein Drink
- Group C: Ice Chips: The control group consisting patient receiving 11 ounces of ice chips
  Interventions: Other: Ice Chips

INTERVENTIONS:
Other: Ice Chips — 11 ounces of ice chips given to the laboring parturient
  Groups: Group C: Ice Chips
Other: Protein Drink — Patients will receive 11 ounces of a protein shake which contains 30 grams of protein
  Other Names: Premier Nutrition Protein Shake (TM)
  Groups: Group P: High Protein Drink

SUMMARY:
Hypothesis: The volume of gastric contents will be the same for a high protein drink versus ice chips as measured by ultrasound at 20 minute intervals for two hours in the laboring parturient.

Specific Aim: To determine the volume of gastric contents at various time intervals (every 20 minutes for 2 hours) in patients with an epidural that are given a high protein drink versus those that are given ice chips, with ultrasound.

DETAILED DESCRIPTION:
Since the 1940s women have had restrictions on oral intake during labor. This idea was first introduced by Mendelson, who raised awareness on the relationship between oral intake during labor and the risk of aspiration of acidic gastric contents if general anesthesia was needed. The aspiration of gastric contents could potentially result in severe maternal morbidity or mortality. As a result, women in labor who receive analgesia are typically restricted to just ice chips in order to prevent aspiration in the rare case that they may require general anesthesia for an emergent or stat cesarean section.

However, recent literature reports that the actual risk of aspiration during labor is extremely low. The risk of aspiration is minimized due to improved general anesthetic techniques involving the use of non-particulate antacids to neutralize gastric acidity and rapid sequence induction to quickly secure the patients airway. Many countries have lenient policies on NPO status during labor, including the Netherlands and United Kingdom, who allow solid food intake during this period.

The policy of "nothing by mouth" during labor and the relationship of aspiration of gastric contents were explored by Mendelson. He experimented on rabbits to explore the effects of gastric contents on their lungs. The rabbits only died when they aspirated material containing hydrochloric acid, and no deaths were due to aspiration of fluids with a neutral pH. Therefore, if oral intake in labor were to be permitted, the ideal characteristics would be for the substance to be in liquid form, isotonic, normothermic, pH of 7.4, and have a low residue.

Labor can be compared to continuous moderate aerobic exercise and these women can experience a state of accelerated starvation. This state of starvation results in the production of ketones for an alternative source of energy. There is much debate about whether this production is harmful to the mother or fetus. A study done by Kubli in 2002 evaluated the effects of isotonic sports drinks and the production of ketones. The drinks decreased ketosis but proved no benefit regarding labor outcome (i.e. length of labor, spontaneous delivery rate). It is important to note that isotonic sports drinks do not contain a significant amount of protein.

It is common for many women in labor to experience nausea and emesis. Protein intake during labor may have a beneficial effect in the prevention of nausea and emesis. The feeling of nausea is experienced when stomach muscles contract irregularly and protein has been shown to re-establish a normal, steadier, and slower rhythm. Protein has been believed to decrease incidence of nausea by decreasing these so-called gastric arrhythmias more so than a carbohydrate meal can (i.e. non-beneficial effect of isotonic sports drinks). It has also been shown that high protein intake decreases nausea and emesis in patients receiving cancer chemotherapy. Furthermore, it has been determined that administration of a protein-rich intake prevents nausea whether given 5 minutes or 45 minutes prior to the nauseating stimuli (i.e. cancer chemotherapy).

It is traditionally thought that gastric emptying in pregnancy is delayed related to changes in hormones such as progesterone as well as the increased abdominal pressure on the gastrum. Perlas et al. has determined that bedside ultrasonography can be a useful non invasive tool to determine gastric content and volume and that the gastric antrum view is the best view to determine gastric volume. In their study of 18 healthy volunteers, a complete cross sectional view of the antrum was obtained 100% of the time, and they found the correlation coefficient to be 0.86 in the right lateral decubitus position. However, their study was not performed on pregnant women.

Wong and colleagues have done several gastric emptying studies after ingestion of water using ultrasound on obese and non-obese non-laboring parturients. In their study of term non laboring women, they found gastric emptying half time was shorter (24 min vs. 33 min) after the ingestion of 300 ml of water than after 50 ml of water. In term obese pregnant women, they did not find any significant difference in gastric emptying after ingestion of 300 ml vs 50 ml. In effect, all water in both studies was back to baseline level at 60 mins post ingestion.

We are unaware of the gastric emptying time of protein solution in pregnant women. Barret et al. has determined that complete gastric emptying of a protein solution takes approximately 2 hours as compared to 1 hour for a glucose solution, and 3 hours for a solid meal in healthy non pregnant adults.

As a follow up to the protein study (PRO10070074), we plan on evaluating the gastric emptying of the protein drink and ice chips using ultrasound to determine gastric volume as described above.

ELIGIBILITY:
Inclusion Criteria:

* All women of childbearing age (including children aged 14 years and above) who request epidural analgesia at Magee-Womens Hospital of UPMC will be eligible to participate in the study
* All participants will be recruited at Magee-Womens Hospital
* All women must present ≤ 5cm cervical dilatation at the time of epidural insertion
* > 36 weeks gestation
* Singleton pregnancy
* Vertex presentation
* NPO ≥ 4 hours prior to epidural insertion

Exclusion Criteria:

* Women with diabetes (at increased risk for gastroparesis and fetal macrosomia)
* Multiple gestation
* Non-vertex fetal presentation
* Chronic opioid use (delayed gastric emptying)
* History of gastric bypass surgery (abnormal anatomical stomach)
* Severe morbid obesity (BMI > 40kg/m2 due to increased intragastric pressure)
* History of known obstetric or medical complication (i.e. preeclampsia) that may increase the likelihood of a complicated or operative delivery (i.e. cesarean section)
* No exclusion criteria shall be based on race and ethnicity
* Men will not be included since they cannot become pregnant

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All women of childbearing age (including children aged 14 years and above) who request epidural analgesia at Magee-Womens Hospital of UPMC will be eligible to participate in the study. The racial, gender and ethnic characteristics of the proposed subject population reflects the demographics of Pittsburgh and the surrounding area and/or the patient population of the University of Pittsburgh Medical Center Health System. Every attempt will be made to recruit subjects in respective proportion to these demographics.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Gastric Emptying | 2 hours
  Gastric emptying will be measured with ultrasounds every twenty minutes for two hours

CONTACTS AND LOCATIONS:
Overall Officials: Manuel C Vallejo, MD, Principal Investigator — Physician Services Division (UPP and CMI) | UPP | Anesthesiology and Pain Medicine
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States